CLINICAL TRIAL: NCT05994235
Title: A Phase II Trial of Tazemetostat Plus Mosunetuzumab in Untreated Follicular Lymphoma
Brief Title: Tazemetostat and Mosunetuzumab in Untreated Follicular Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Epizyme, Inc. (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-06026184; 22-10025285 (Other: WCM IRB)
Record Dates: First submitted 2023-08-08; First posted 2023-08-16 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Follicular Lymphoma
Keywords: Mosunetuzumab; Follicular Lymphoma; Tazemetostat
MeSH Terms: conditions — Lymphoma, Follicular | interventions — tazemetostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Subcutaneous Mosunetuzumab and Oral Tazemetostat (Experimental): 50 patients will be enrolled and treated with standard dosing of subcutaneous mosunetuzumab, and with oral tazemetostat by mouth twice daily at standard dosing (800 mg twice daily) beginning at the same time as mosunetuzumab initiation.
  Interventions: Drug: Mosunetuzumab; Drug: Tazemetostat Pill

INTERVENTIONS:
Drug: Mosunetuzumab — Mosunetuzumab will be administered in weekly dose increments ("step-up dosing") during Cycle 1 and then on Day 1 of each cycle. Mosunetuzumab will be given in 28-day cycles for up to 12 cycles. Mosunetuzumab will be administered SC at the dose of 5 mg on Day 1, 45 mg on Day 8, and 45 mg on Day 15 in Cycle 1. Beginning with Cycle 2, it will be administered SC at the dose of 45 mg on Day 1. Each cycle lasts 4 weeks.
Drug: Tazemetostat Pill — Oral tazemetostat will be administered by mouth twice daily at standard dosing (800 mg twice daily) beginning at the same time as mosunetuzumab initiation until disease progression, unacceptable toxicity, or consent is withdrawn. Patients will remain on tazemetostat for up to twelve 28-day cycles from initiation of mosunetuzumab.
  Other Names: Tazverik

SUMMARY:
The goal of this study is to learn about the safety and effectiveness of the combination of tazemetostat pills in combination with mosunetuzumab injections for people with follicular lymphoma who haven't received treatment before. The investigators hypothesize that tazemetostat with mosunetuzumab has the potential to increase the efficacy of the product without compromising the safety.

Tazemetostat is a drug that inhibits EZH2, an enzyme known to drive the development of B-cell lymphomas, and inhibiting it appears to have many effects that slow down lymphoma growth and enhance the immune system's ability to fight it. Tazemetostat is FDA-approved in previously treated follicular lymphoma and currently undergoing study in other lymphomas.

Mosunetuzumab is a bispecific antibody therapy that is a therapeutic strategy that uses the immune system to fight lymphoma, called immunotherapy. Bispecific antibodies have two ends: one attaches to T cells in the immune system and the other attaches to lymphoma cells, helping guide our immune system to attack the cancer. Mosunetuzumab has been studied in follicular lymphoma that has previously been treated, with positive results. Mosunetuzumab is approved by the FDA to be given intravenously (directly into a vein) but is not yet approved by the FDA is not yet approved as an injection under the skin, which is how it is given in this study. They have not yet been studied in combination.

DETAILED DESCRIPTION:
This is a phase II, open-label study. Fifty patients will be enrolled and treated with standard dosing of SC mosunetuzumab, and with oral tazemetostat by mouth twice daily at standard dosing (800 mg twice daily) beginning at the same time as mosunetuzumab initiation. Response assessments by PET/CT will occur post-mosunetuzumab at Cycle 4, Day 1 (+/- 3 days) and again at the end of treatment. If a participant has a complete response (CR) at Cycle 4 and/or cycle 8, then they will receive a total of 8 cycles of mosunetuzumab. If the patient has a partial response or stable disease at Cycle 4 and Cycle 8, then they will receive a total of 12 cycles of mosunetuzumab. All participants will receive 12 cycles of tazemetostat, unless discontinued from treatment early for disease progression or other protocol-defined reasons. Treatment with steroids, tocilizumab, growth factors, tumor lysis prophylaxis, and antibiotics may be used as per standard of care at our institution. Dose modifications are permitted for toxicity. Correlative studies will be performed prior to and following tazemetostat treatment and peripheral blood collections prior to post-mosunetuzumab treatment, which will give additional descriptive data for use in correlative analyses.

ELIGIBILITY:
Inclusion Criteria

Patients must meet the following criteria for study entry:

* Signed Informed Consent Form
* Age: 18 years at the time of signing the Informed Consent Form
* Ability to comply with the study protocol
* Willing to follow lifestyle considerations as defined in Section 4.4
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1, or 2
* Histologically documented FL (Grades 1-3a):

  * Fluorodeoxyglucose avid lymphoma (i.e., positron emission tomography (PET) positive lymphoma)
  * At least 1 bi-dimensionally measurable nodal lesion (˃1.5 cm in its largest dimension by computed tomography (CT) scan), or at least 1 bi-dimensionally measurable extra-nodal lesion (˃1.0 cm in its largest dimension by CT scan)
* Meet Groupe d'Etude des Lymphomes Folliculaires (GELF) criteria to receive systemic therapy
* Received no prior systemic lymphoma therapy (local radiotherapy is not considered systemic therapy)
* Availability of a representative tumor specimen and the corresponding pathology report at the time of diagnosis for confirmation of the diagnosis of FL and for EZH2 mutation testing.
* Adequate hematologic function defined as follows:

  * Hemoglobin >= 8.0 g/dL
  * ANC >=1.0 x 10/L
  * Platelet count >=75x10/L
* Adequate renal and hepatic function as defined as follows:

  * Measured or estimated creatinine clearance >=30 mL/min by institutional standard method
  * AST or ALT <= 2.5 x the upper limit of normal (ULN)
  * Serum total bilirubin <=1.5xULN (or <=3 x ULN for patients with Gilbert syndrome)

Patients who meet any of the following criteria will be excluded from study entry:

* Inability to take oral medication OR have malabsorption syndrome or any other uncontrolled gastrointestinal condition (eg, nausea, diarrhea, vomiting) that might impair the bioavailability of tazemetostat
* Grade 3b FL
* History of transformation of indolent disease to diffuse large B cell lymphoma
* Any prior history of myeloid malignancies, including myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML) or myeloproliferative neoplasm (MPN)
* Any prior history of T-LBL/T-ALL
* Active or history of CNS lymphoma or leptomeningeal infiltration
* Prior standard or investigational systemic anti-cancer therapy for lymphoma. Patients who have received prior XRT will not be excluded
* Treatment with systemic immunosuppressive medications, including, but not limited to, prednisone (20 mg), azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor agents within 2 weeks prior to Day 1 of Cycle 1

  * The use of inhaled corticosteroids is permitted
  * The use of mineralocorticoids for the management of orthostatic hypotension is permitted
  * Dexamethasone for nausea, B symptoms, or symptomatic or bulky disease is permitted with a maximum dose of 40 mg x5 days or equivalent
* History of solid organ transplantation
* Contraindication to tocilizumab
* History of severe allergic or anaphylactic reaction to humanized, chimeric or murine monoclonal antibodies (MAbs)
* Known hypersensitivity to biopharmaceuticals produced in CHO cells or any component of the mosunetuzumab or tazemetostat.
* Known active bacterial, viral, fungal, or other infection, or any major episode of infection requiring treatment with IV antibiotics within 4 weeks of Day 1 of Cycle 1
* Known or suspected chronic active Epstein-Barr virus (EBV) infection
* Known or suspected history of hemophagocytic lymphohistiocytosis (HLH)
* Clinically significant history of liver disease, including viral or other hepatitis, or cirrhosis, as determined by the principal investigator
* Active Hepatitis B or Hepatitis C infection Note: Patients who are hepatitis B surface antigen (HBsAg) negative and hepatitis B core antibody (HBcAb) positive, must be negative for hepatitis B virus (HBV) polymerase chain reaction (PCR) to be eligible for study participation. Patients who are positive for hepatitis C virus (HCV) antibody must be negative for HCV by PCR to be eligible for study participation
* HIV positive with CD4 count <200 and not currently taking antiretroviral therapy
* History of progressive multifocal leukoencephalopathy (PML)
* Administration of a live, attenuated vaccine within 4 weeks before first dose of study treatment or anticipation that such a live attenuated vaccine will be required during the study

  * Patients must not receive live, attenuated vaccines (e.g., FluMist) while receiving study treatment or after the last dose until B-cell recovery to the normal ranges.
  * Inactivated influenza vaccination should be given during the influenza season only
* Other malignancy that could affect compliance with the protocol or interpretation of results, with the exception of the following:

  * Any of the following malignancies previously curatively treated: carcinoma in situ of the cervix, good-prognosis ductal carcinoma in situ of the breast, basal, or squamous cell skin cancer
  * Stage I melanoma, - Low-grade, early-stage localized prostate cancer
  * Any other previously treated malignancy that has been in remission without treatment for >= 2 years prior to enrollment
* Active autoimmune disease requiring treatment
* History of autoimmune disease, including, but not limited to: myocarditis, pneumonitis, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis

  * Patients with a remote history of, or well-controlled autoimmune disease, with a treatment free interval from immunosuppressive therapy for 12 months may be eligible to enroll if judged to be safe by the investigator
  * Patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid-replacement hormone are eligible Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study
  * Patients with a history of disease-related immune thrombocytopenic purpura, or autoimmune hemolytic anemia may be eligible
* Prior allogeneic stem cell transplant (SCT)
* Evidence of any significant, uncontrolled concomitant disease that could affect compliance with the protocol or interpretation of results, including, but not limited to, significant cardiovascular disease (e.g., New York Heart Association Class III or IV cardiac disease, myocardial infarction within the previous 6 months, unstable arrhythmia, or unstable angina) or significant pulmonary disease (such as obstructive pulmonary disease or history of bronchospasm)
* Major surgical procedure other than for diagnosis within 28 days prior to Day 1 of Cycle 1 Day 1 or anticipation of a major surgical procedure during the course of the study
* Active CNS disease or underlying neurologic disease such as stroke or intracranial hemorrhage within 3 months prior to enrollment, history of seizure disorder, or history of neurogenerative disease
* History of pneumonitis or interstitial lung disease
* A positive SARS-CoV-2 test within 7 days of C1D1
* Pregnant or lactating or intending to become pregnant during the study

  * Women of childbearing potential (WOCBP) must have 2 negative serum pregnancy test results (minimum sensitivity, 25 mIU/mL) prior to initiating therapy: at 10-14 days prior to Day 1 of Cycle 1 and within 24 hours prior to Day 1 of Cycle 1.
  * WOCBP are defined as any person with a uterus who has had a menstrual period in the last 12 months, unless surgically sterile (i.e. from hysterectomy or bilateral oophorectomy)
* Any serious medical condition or abnormality in clinical laboratory tests that, in the investigator's judgment, precludes the patient's safe participation in and completion of the study, or which could affect compliance with the protocol or interpretation of results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2033-10 (Estimated); Study Completion 2033-10 (Estimated)

PRIMARY OUTCOMES:
Number of participants who achieve a complete response (CR) by completion of therapy, as determined by the Lugano Criteria | Estimated day 336
  The proportion of patients who achieve complete response as per the Lugano criteria will be calculated and their 90% confidences will be computed with Clopper-Pearson method via exact binomial distribution.

SECONDARY OUTCOMES:
Number of participants who experience cytokine release syndrome (CRS) | Day 0 to Day 28
  CRS will be assessed per American Society for Transplantation and Cellular Therapy (ASTCT) Consensus Grading
Number of participants who experience Immune effector cell-associated neurotoxicity syndrome (ICANS) | Day 0 to Day 28
  ICANS will be assessed per American Society for Transplantation and Cellular Therapy (ASTCT) Consensus Grading
Median Progression-Free Survival (PFS) | For a maximum of approximately 10 years
  PFS is defined as the duration of time from start of treatment to time of progression or death from any cause. Patients will be followed for a maximum of approximately 10 years from the start of treatment.
Median Overall Survival (OS) | For a maximum of approximately 10 years
  OS is defined as the duration of time from start of treatment to death from any cause. Patients will be followed for a maximum of approximately 10 years from the start of treatment.
Objective Response Rate (ORR) at the time of therapy completion, as defined by Lugano Criteria | Estimated to be day 336
  ORR is defined as the proportion of patients who have a partial or complete response to therapy
Number of participants who achieve a Complete Response (CR) per Lugano's Criteria | For a maximum of approximately 10 years
  Response and progression are evaluated according to the Lugano criteria for lymphoma response.
Median Duration of Response | For a maximum of approximately 10 years
  The duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease or death due to any cause, whichever occurs first is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started).

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Yamshon, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine/NewYork-Presbyterian Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No